CLINICAL TRIAL: NCT00441181
Title: Effects of Travoprost on Neovascular Glaucoma
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UNIFESP 2007-02
Record Dates: First submitted 2007-02-27; First posted 2007-02-28 (Estimated); Last update posted 2011-06-22 (Estimated); Status verified 2007-02

CONDITIONS: Neovascular Glaucoma
Keywords: Neovascular glaucoma; Travoprost
MeSH Terms: conditions — Glaucoma, Neovascular | interventions — Travoprost

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Travoprost

SUMMARY:
Prostaglandin analogues have not been used in the treatment of neovascular glaucoma because of suspicious lack of efficacy. This study aims at assessing the effect of travoprost on neovascular glaucoma.

ELIGIBILITY:
Inclusion Criteria:

* Neovascular glaucoma of known cause
* Older than 18 years
* Previously submitted to retinal photocoagulation
* Under medical treatment to glaucoma

Exclusion Criteria:

* Need of antiglaucomatous surgery
* Previous ocular surgery in the last 6 months
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2008-01; Study Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
Intraocular pressure

SECONDARY OUTCOMES:
Inflammation

CONTACTS AND LOCATIONS:
Overall Officials: Luiz A Melo Jr, MD, Principal Investigator — Federal University of São Paulo
Locations (1):
- Federal University of São Paulo, São Paulo, São Paulo, Brazil